CLINICAL TRIAL: NCT01416480
Title: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of "Theobromine Capsule 300mg" as an Antitussive Agent in Acute Cough Patients.
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of "Theobromine Capsule" as an Antitussive in Acute Cougher
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Jung Hoon, Han / Senior Researcher, Project Development Team / Ahn-Gook Pharmaceuticals Co.,Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG1321001_ACP3
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Acute Bronchitis
Keywords: Theobromine; cough; acute bronchitis
MeSH Terms: conditions — Bronchitis; Cough | interventions — Theobromine; dipropizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theobromine (Experimental): Theobromine capsule 300mg
  Interventions: Drug: Theobromine 300mg
- levodropropizine (Active Comparator): levodropropizine syrup
  Interventions: Drug: Levodropropizine 10mg

INTERVENTIONS:
Drug: Theobromine 300mg — Capsule, b.i.d.
  Arms: Theobromine
Drug: Levodropropizine 10mg — Syrup, t.i.d.
  Arms: levodropropizine

SUMMARY:
The aim of this clinical trial is to evaluate the antitussive effect of "Theobromine capsule 300mg" in patients with acute bronchitis.

DETAILED DESCRIPTION:
This study is double blinded, randomized, parallel designed, phase III clinical trial to evaluate the efficacy and safety of "Theobromine capsule 300mg" versus "Levodropropizine syrup" in patients with acute bronchitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who decided to participate in this clinical trial at his(her) own will and agreed in written letter of consent.
2. Adult aged over 18
3. Patient who has cough symptom caused by acute bronchitis
4. Patient who go to see the doctor for severe cough at his(her) own will
5. DCS score at screening vist sould be over 3.
6. For fertile woman, HCG test at screening visit shloud be negative.

patient who will continue to cough more than 1 week.(by physician's judgment)

Exclusion Criteria:

1. Patient who is accompanied by the seriously abnormal symptom in respiratory system, such as Acute infectious Pulmonary Disease, Tuberculosis, asthma.
2. Chronic bronchitis including bronchial obstruction
3. Patient who has clinical history of sensitivity to Xanthine drug.
4. Patient who has Peptic Ulcer
5. Patient whose liver or kidney function is seriously abnormal: Including the cases of sGOT, sGPT, bilirubin and blood creatinine value exceeding twice of their upper normal limit.
6. Patient whose heart function is abnormal: including the case of showing abnormal EKG test value that is clinically significant.
7. patient who has convulsion or alcoholism.
8. Patient who has experience to have participated in other clinical trial within two months before starting the trial.
9. Pregnant woman, lactating woman.
10. Patient who thought to be cured within 3 days without any medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
cough remission rate | 3 days
  cough remission : no cough or 1 short cough in day time

SECONDARY OUTCOMES:
cough recovery rate | 1 day, 2 days, within 3days
difference of DCS score between screening and closing visit. | 3 days
required time for cough remission | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Suck Jung, M.D., Principal Investigator — Hallym University Medical Center; Soo-Taek Uh, M.D., Principal Investigator — Soon Chun Hyang University Hospital; Jae Yeol Kim, M.D., Principal Investigator — Chung-Ang University Medical Center; Young Kyoon Kim, M.D., Principal Investigator — The Catholic University of Korea-St. Mary's Hospital; Sung Soon Lee, M.D., Principal Investigator — Inje University Ilsan Paik Hospital; Yong Bum Park, M.D., Principal Investigator — Kangdong Sacred Heart Hospital; Kwan Ho Lee, M.D., Principal Investigator — Yeungnam University Hospital; Jung Hyun chang, M.D., Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Hallym University Medical Center, Anyang-si, Gyeonggi-do, South Korea